CLINICAL TRIAL: NCT02519322
Title: Neoadjuvant and Adjuvant Checkpoint Blockade in Patients With Clinical Stage III or Oligometastatic Stage IV Melanoma
Brief Title: Neoadjuvant and Adjuvant Checkpoint Blockade
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0041; NCI-2015-01520 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0041 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cutaneous Melanoma; Mucosal Melanoma; Ocular Melanoma; Stage III Acral Lentiginous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIB Uveal Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IIIC Uveal Melanoma AJCC v7; Stage IV Acral Lentiginous Melanoma AJCC v6 and v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; relatlimab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (nivolumab, surgery) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1, 15, 29, and 43. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery
- Arm B (nivolumab, ipilimumab, surgery) (Experimental): Patients receive nivolumab IV over 1 hour and ipilimumab IV over 90 minutes on days 1, 22, and 43. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery
- Arm C (nivolumab, relatlimab, surgery) (Experimental): Patients receive nivolumab IV over 1 hour and relatlimab IV over 1 hour on days 1 and 29. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 1 hour and relatlimab IV over 1 hour every 4 weeks for 10 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Biological: Relatlimab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm B (nivolumab, ipilimumab, surgery)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Relatlimab — Given IV
  Other Names: BMS-986016; BMS986016; Immunoglobulin G4, Anti-(human Lymphocyte Activation Gene-3 Protein) (Human Heavy Chain), Disulfide with Human Light Chain, Dimer
  Arms: Arm C (nivolumab, relatlimab, surgery)
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This randomized phase II trial studies how well nivolumab with or without ipilimumab or relatlimab before surgery works in treating patients with stage IIIB-IV melanoma that can be removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab, ipilimumab, and relatlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving nivolumab alone or in combination with ipilimumab or relatlimab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pathologic response of nivolumab monotherapy and nivolumab and ipilimumab dual therapy administered in the neoadjuvant setting in patients with high-risk resectable melanoma. Pathologic response will be assessed by percent viable tumor cells, percent tumor necrosis, presence of fibrosis and melanoma proliferation as assessed by phosphohistone H3 from baseline, to on-treatment and surgical specimens. (Arm A and Arm B) II. To assess the pathologic response rate of combination relatlimab with nivolumab in the neoadjuvant setting in patients with high-risk resectable Stage IIIB/C or oligometastatic Stage IV melanoma. Pathologic response will be assessed by percent viable tumor cells, percent tumor necrosis, presence of fibrosis and melanoma proliferation as assessed by phosphohistone H3 from baseline, to on- treatment and surgical specimens. (Arm C)

SECONDARY OBJECTIVES:

I. To assess the immunologic response of neoadjuvant nivolumab monotherapy and neoadjuvant nivolumab and ipilimumab dual therapy in patients with high-risk resectable melanoma. Immunologic response will be determined by change in T cell infiltrate from baseline to on-treatment and surgical specimens in response to therapy. (Arm A and Arm B) II. To assess the objective response rate (ORR) of nivolumab monotherapy and nivolumab and ipilimumab dual therapy administered in the neoadjuvant setting as assessed by imaging (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) in patients with high-risk resectable melanoma. (Arm A and Arm B) III. To assess the 12-month recurrence-free survival (RFS) and overall survival (OS) of patients with high-risk resectable melanoma treated with neoadjuvant nivolumab monotherapy or nivolumab and ipilimumab dual therapy followed by adjuvant nivolumab. (Arm A and Arm B) IV. To evaluate the safety of nivolumab monotherapy and dual ipilimumab and nivolumab in the neoadjuvant setting and peri-operatively as well as assess the safety of adjuvant nivolumab. (Arm A and Arm B) V. To evaluate safety and feasibility of relatlimab with nivolumab delivered in the neoadjuvant setting. (Arm C) VI. To assess the objective response rate (ORR) of relatlimab with nivolumab administered in the neoadjuvant setting as assessed by imaging (RECIST 1.1 criteria) in patients with high-risk resectable melanoma. (Arm C) VII. To assess the 12-month recurrence-free survival (RFS) and overall survival (OS) of patients with high-risk resectable melanoma treated with neoadjuvant and adjuvant relatlimab with nivolumab. (Arm C) VIII. To evaluate immunologic and molecular mechanisms of response and resistance to relatlimab with nivolumab. (Arm C)

EXPLORATORY OBJECTIVES:

I. Identification of immunologic and genomic markers correlating with clinical response or resistance to nivolumab monotherapy and ipilimumab with nivolumab combination therapy.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes on days 1, 15, 29, and 43. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity. (CLOSED TO ENROLLMENT AS OF 10/3/2018)

ARM B: Patients receive nivolumab IV over 1 hour and ipilimumab IV over 90 minutes on days 1, 22, and 43. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity. (CLOSED TO ENROLLMENT AS OF 10/3/2018)

ARM C: Patients receive nivolumab IV over 1 hour and relatlimab IV over 1 hour on days 1 and 29. Patients then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 1 hour and relatlimab IV over 1 hour every 4 weeks for 10 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Patients must have histologically or cytologically confirmed stage IIIB/C or stage IV oligometastatic melanoma; oligometastatic melanoma is defined as three or fewer areas of resectable disease excluding central nervous system and bone involvement; patients with cutaneous, mucosal, acral, ocular or unknown primary melanomas are eligible for enrollment; for patients with stage IV disease with distant lymph nodes (stage M1a), a maximum of three separate lymph node sites fit the definition of oligometastatic disease; resectable tumors are defined as having no significant vascular, neural or bony involvement; only cases where a complete surgical resection with tumor-free margins can safely be achieved are defined as resectable
* Patients will have at least one melanoma deposit that can undergo serial biopsy (at least 2 time points) during the neoadjuvant phase of the protocol; patients must be willing to provide tumor samples at the time points specified in the Study Procedure Tables
* All patients must undergo a baseline tumor biopsy; in Arms A and B, tumor biopsy for PD-L1 testing (PD-L1 positivity is determined by greater than or equal to 1% of cells staining in the membrane by immunohistochemistry) is required for stratification; PD-L1 status is not required for enrollment on Arm C; the 28-8 clone for PD-L1 testing is required for assessment of PD-L1 status; for patients with stage IV disease, site of tumor biopsy will preferably be from non-lymph node disease site; for PD-L1 testing, the biopsy should contain sufficient tumor content (> 100 tumor cells/4-micron tissue section); if a sample contains insufficient tumor content, a re-biopsy will be required to obtain a sample with sufficient tumor content prior to treatment
* Patients must be medically fit enough to undergo surgery as determined by the treating medical and surgical oncology team
* Patients who have been previously treated in the adjuvant setting for melanoma will be eligible for treatment after a 28 day wash-out period
* Patients must have measurable disease, defined by RECIST 1.1
* Age >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L (within 28 days of first study treatment)
* Hemoglobin >= 8.5 g/dL (within 28 days of first study treatment)
* Platelets >= 100 X 10^9/L (>= 60 for hepatocellular carcinoma [HCC]) (within 28 days of first study treatment)
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 X upper limit of normal (ULN) (within 28 days of first study treatment)
* White blood cells (WBC) >= 2.0 X 10^9/L (within 28 days of first study treatment)
* Total bilirubin =< 1.5 X ULN (except subjects with Gilbert's syndrome who must have normal direct bilirubin) [3 mg/dL for HCC] (within 28 days of first study treatment)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x upper limit of normal (ULN) (=< 5 x ULN for HCC) (within 28 days of first study treatment)
* Albumin >= 2.5 g/dL (within 28 days of first study treatment)
* Creatinine =< 1.5 x ULN OR calculated creatinine clearance >= 40 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min (within 28 days of first study treatment)
* Lipase < 1.5 X ULN (within 28 days of first study treatment)
* Amylase < 1.5 X ULN (within 28 days of first study treatment)
* Normal thyroid function (or stable on hormone supplementation) 0.27 - 10 X 10^9/L (within 28 days of first study treatment)
* Left ventricular ejection fraction (LVEF) >= 50% by transthoracic echocardiography (TTE) (preferred) or multigated acquisition (MUGA) within 6 months from first study drug administration
* Women are eligible to participate if: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] > 40 MlU/mL and estradiol < 40 pg/mL [< 140 pmol/L] is confirmatory); females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study; otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment; for most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT; following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* A woman of childbearing potential (WOCBP) agrees to use method(s) of contraception; for a teratogenic study drug and/or when there is insufficient information to assess teratogenicity, a highly effective method(s) of contraception (failure rate of < 1% per year) is required; the individual methods of contraception and duration should be determined in consultation with the investigator; WOCBP must follow instructions for birth control when the half-life of the study drug is > 24 hours; contraception should be continued for a period of 30 days plus the time required for the study drug to undergo 5 half-lives; WOCBP should use an adequate method to avoid pregnancy for 24 weeks (30 days plus the time required for study drug to undergo 5 half-lives) after the last dose of study drug; WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of investigational product
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of < 1% per year; the investigator shall review contraception methods and the time period that contraception must be followed; men who are sexually active with WOCBP must follow instructions for birth control when the half-life of the study drug is > 24 hours, contraception should be continued for 90 days plus the time required for the study drug to undergo 5 half-lives; therefore, men who are sexually active with WOCBP must continue contraception for 33 weeks (90 days plus the time required for nivolumab and/or relatlimab to undergo 5 half-lives) after the last dose of study drug; in addition, male participants must be willing to refrain from sperm donation during this time; men who are sexually active with women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile and azoospermic men) do not require contraception
* For Arm C: Cardiac assessment at baseline by trans- thoracic echocardiogram (TTE) with LVEF 50%

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug
* Any major surgery within the last 3 weeks
* Brain metastases, leptomeningeal disease or bone metastases
* Pregnant or lactating female
* Unwillingness or inability to follow the procedures required in the protocol
* Current use of anticoagulants (warfarin, heparin, direct thrombin inhibitors) at therapeutic levels
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Prior malignancy active within the previous 3 years except for patient's prior diagnosis of melanoma and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast with local control measures (surgery, radiation)
* Subjects with active, known or suspected autoimmune disease; subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-LAG-3, or anti-CTLA-4 antibody
* Any positive test result for hepatitis B or C virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of severe hypersensitivity reaction to any monoclonal antibody
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (infection disease) illness
* A known or underlying medical condition that, in the opinion of the Investigator, could make the administration of the study drug hazardous to the subject or could adversely affect the ability of the subject to comply with or tolerate the study
* A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
* Evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy 7 days prior to initiation of study drug therapy
* Any other acute or chronic medical illness
* Subjects who are unable to undergo venipuncture and/or tolerate venous access
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator
* Any of the following procedures or medications:

  * Within 2 weeks prior to time of study treatment:

    * Systemic or topical corticosteroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent); inhaled or topical steroids, and adrenal replacement steroid doses of > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
    * Palliative radiation or gamma
  * Within 4 weeks prior to study drug administration:

    * Any investigational cytotoxic drug; exposure to any non-cytotoxic drug within 4 weeks or 5 half-lives (whichever is shorter) is prohibited; if 5 half-lives is shorter than 4 weeks, agreement with sponsor/medical monitor is mandatory
* Subjects with history of life-threatening toxicity related to prior immune therapy (e.g., anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (e.g., hormone replacement after endocrinopathy)
* Troponin T (TnT) or I (TnI) > 2 x institutional upper limit of normal (ULN); subjects with TnT or TnI levels between > 1 to 2 x ULN will be permitted if repeat levels within 24 hours are </= 1 x ULN; if TnT or TnI levels are > 1 to 2 x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the investigator or designee; when repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible; if TnT or TnI repeat levels beyond 24 hours are < 2 x ULN, the subject may undergo a cardiac evaluation and be considered for treatment, following a discussion with the investigator or designee
* For Arm C: Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
  * Uncontrolled angina within the 3 months prior to consent
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * Corrected QT interval (QTc) prolongation > 480 msec
  * History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, deep venous thrombosis, etc )
  * Cardiovascular disease-related requirement for daily supplemental oxygen
  * History of two or more MIs OR two or more coronary revascularization procedures
  * Subjects with history of myocarditis, regardless of etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Burton EM, Milton DR, Tetzlaff MT, Wani K, Ross MI, Postow MA, Lazcano R, Glitza IC, Wong MK, Patel SP, Diab A, Gershenwald JE, McQuade JL, Betof Warner A, Prieto VG, Lee JE, Goepfert RP, Fisher SB, Song A, Malke J, Simon JM, Ariyan C, Torres-Cabala CA, Davies MA, Lazar A, Wargo JA, Tawbi HA, Amaria RN. Long-Term Survival and Biomarker Analysis Evaluating Neoadjuvant Plus Adjuvant Relatlimab (anti-LAG3) and Nivolumab (anti-PD1) in Patients With Resectable Melanoma. J Clin Oncol. 2025 Sep 10;43(26):2856-2862. doi: 10.1200/JCO-25-00494. Epub 2025 Jul 10. PMID 40638872
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized non-comparative sugy of neoadjuvant nivolumab monothereapy or nivolumab combined with ipilimumab followed by adjuvant nivolumab or nivolumabe combined with relatlimab in adult (> 18 years) subjects with resectable, high-risk melanoma.
Pre-assignment Details: The number of participants enrolled were 53. However, data was not captured for 19 participants in Arms A & B. 34 participants in Arm C were treated.
Groups:
- Arm A (Nivolumab, Surgery): Participants receive nivolumab IV over 30 minutes on days 1, 15, 29, and 43. Participants then undergo surgery on day 57. After surgery, patients receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
- Arm B (Nivolumab, Ipilimumab, Surgery): Participants receive nivolumab IV over 1 hour and ipilimumab IV over 90 minutes on days 1, 22, and 43. Patients then undergo surgery on day 57. After surgery, Participants receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
- Arm C (Nivolumab, Relatlimab, Surgery): Participants receive nivolumab IV over 1 hour and relatlimab IV over 1 hour on days 1 and 29. Participants then undergo surgery on day 57. After surgery, Participants receive nivolumab IV over 1 hour and relatlimab IV over 1 hour every 4 weeks for 10 doses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Relatlimab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
Period: Overall Study
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Started | 0 | 0 | 34
Completed | 0 | 0 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were in the Arm A or Arm B only Arm C
Groups:
- Arm A (Nivolumab, Surgery): Nivolumab IV over 30 minutes D1, 15, 29, & 43; Surgery D57; Post-surgery Nivolumab IV over 30 minutes Q2wks for 13 doses
- Arm B (Nivolumab, Ipilimumab, Surgery): Nivolumab IV ocer 1 hr and ipilimumab IV over 90 minutes D1, 22, & 43; Surgery D57; Nivolumab IV over 30 minutes Q2wks for 13 doses
- Arm C (Nivolumab, Relatlimab, Surgery): Nivolumab IV and relatilmab IV over 1 hr D1 and D29; Surgery D57; Post-surgery Nivolumab IV and relatimab IV over 1 hr Q4wks for 10 doses
- Total: Total of all reporting groups
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery) | Total
Number analyzed (Participants) | 0 | 0 | 34 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 23 | 23
  >=65 years |  |  | 11 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 13 | 13
  Male |  |  | 21 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 2 | 2
  Not Hispanic or Latino |  |  | 24 | 24
  Unknown or Not Reported |  |  | 8 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0
  Asian |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0
  Black or African American |  |  | 0 | 0
  White |  |  | 32 | 32
  More than one race |  |  | 0 | 0
  Unknown or Not Reported |  |  | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States |  |  | 34 | 34

OUTCOME MEASURES:

1. Primary Outcome: Arm C: Number of Participants With the Pathologic Response Rate
Description: Number of participants with the Pathologic response rate will be assessed by percent viable tumor cells, percent tumor necrosis, presence of fibrosis and melanoma proliferation as assessed by phosphohistone H3 from baseline, to on-treatment and surgical specimens.
Time Frame: up to 2 years
Population: No data to report due to study Closed to entry as of 07/2017 regarding Arm A and Arm B.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Nivolumab, Surgery): Participants receive nivolumab IV over 30 minutes on days 1, 15, 29, and 43. Participants then undergo surgery on day 57. After surgery, participants receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
- Arm B (Nivolumab, Ipilimumab, Surgery): Participants receive nivolumab IV over 1 hour and ipilimumab IV over 90 minutes on days 1, 22, and 43. Participants then undergo surgery on day 57. After surgery, participants receive nivolumab IV over 30 minutes every 2 weeks for 13 doses in the absence of disease progression or unacceptable toxicity.
  Ipilimumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Number analyzed (Participants) | 0 | 0 | 34
Participants | 0 | 0 | 34

2. Secondary Outcome: Arm C: Number of Participants Assessed by Safety and Feasibility of Relatlimab With Nivolumab Delivered in the Neoadjuvant Setting
Description: Number of Participants assessed by the safety and feasibility of relatlimab with nivolumab Delivered in the Neoadjuvant Setting
Time Frame: up to 2 years
Population: No data to report due to study Closed to entry as of 07/2017 regarding Arm A and Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Number analyzed (Participants) | 0 | 0 | 34
Participants | 0 | 0 | 34

3. Secondary Outcome: Arm C: Number of Participants With Objective Response Rate (ORR) of Relatlimab With Nivolumab Administered in the Neoadjuvant Setting.
Description: To assess the objective response rate (ORR) of relatlimab with nivolumab administered in the neoadjuvant setting as assessed by imaging (RECIST 1.1 criteria) in participants with high-risk resectable melanoma
Time Frame: Up to 2 years
Population: No data to report due to study Closed to entry as of 07/2017 regarding Arm A and Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Number analyzed (Participants) | 0 | 0 | 34
Participants | 0 | 0 | 34

4. Secondary Outcome: Arm C: Number of Participants With Recurrence-Free Survival (RFS) and Overall Survival (OS)
Description: To assess the 12-month recurrence and overall survival (OS) of participants with high-risk resectable melanoma treated with neoadjuvant and adjuvant relatlimab with nivolumab
Time Frame: up to 12 months
Population: No data to report due to study Closed to entry as of 07/2017 regarding Arm A and Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Number analyzed (Participants) | 0 | 0 | 34
Participants | 0 | 0 | 34

5. Secondary Outcome: Arm C: Number of Participants With Immunologic and Molecular Mechanisms of Response and Resistance.
Description: To assess by immunologic and molecular mechanisms of response and resistance to relatlimab with nivolumab.
Time Frame: up to 2 years
Population: No data to report due to study Closed to entry as of 07/2017 regarding Arm A and Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
Number analyzed (Participants) | 0 | 0 | 34
Participants | 0 | 0 | 34

ADVERSE EVENTS:
Time Frame: Baseline to 2 years post treatment
Description: No participants were analyzed in Arm A and Arm B, only in Arm C.
Groups:
- Arm A (Nivolumab, Surgery): Nivolumab IV over 30 minutes D1, 15, 29 & 43; surgery D57; post-surgery nivolumab IV over 30 minutes for Q2wks for 13 doses
- Arm C (Nivolumab, Relatlimab, Surgery): Nivolumab IV ocer 1 hr and ipilimumab IV over 90 minutes D1, 22, & 43; Surgery D57; Nivolumab IV over 30 minutes Q2wks for 13 doses
  Relatlimab: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
Arm/Group | Arm A (Nivolumab, Surgery) | Arm B (Nivolumab, Ipilimumab, Surgery) | Arm C (Nivolumab, Relatlimab, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/34
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 34/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A (Nivolumab, Surgery) (N=0) | Arm B (Nivolumab, Ipilimumab, Surgery) (N=0) | Arm C (Nivolumab, Relatlimab, Surgery) (N=34)
Abdominal Pain (Gastrointestinal disorders) | NA | NA | 4 (6)
Activated partial thromboplastin time prolonged (Investigations) | NA | NA | 2 (2)
Acute kidney injury (Renal and urinary disorders) | NA | NA | 2/33
Adrenal insufficiency (Endocrine disorders) | NA | NA | 8 (11)
Agitation (Psychiatric disorders) | NA | NA | 2
Alanine aminotransferase increased (Investigations) | NA | NA | 14 (23)
Alkaline phosphatase increased (Investigations) | NA | NA | 7 (14)
Alopecia (Skin and subcutaneous tissue disorders) | NA | NA | 2
Anemia (Blood and lymphatic system disorders) | NA | NA | 20 (37)
Anorexia (Metabolism and nutrition disorders) | NA | NA | 9 (11)
Anxiety (Investigations) | NA | NA | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | 10 (16)
Aspartate aminotransferase increased (Investigations) | NA | NA | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | NA | NA | 7 (7)
Bloating (Gastrointestinal disorders) | NA | NA | 2 (2)
Ischemia (Blood and lymphatic system disorders) | NA | NA | 2
Blood bilirubin increased (Investigations) | NA | NA | 5 (6)
Blurred Vision (Eye disorders) | NA | NA | 7 (8)
Bruising (Injury, poisoning and procedural complications) | NA | NA | 2 (2)
Mitral Valve Prolapse (Cardiac disorders) | NA | NA | 2
Tropinin T Increased (Cardiac disorders) | NA | NA | 10 (18)
Hemoptsis (Cardiac disorders) | NA | NA | 2
Tropinin I increased (Cardiac disorders) | NA | NA | 3 (3)
Chills (General disorders) | NA | NA | 6
Colitis (Gastrointestinal disorders) | NA | NA | 3 (5)
Concentration impairment (Nervous system disorders) | NA | NA | 2
Confusion (Nervous system disorders) | NA | NA | 2
Constipation (Gastrointestinal disorders) | NA | NA | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | 18 (23)
CPK increased (Investigations) | NA | NA | 2 (5)
Creatinine increased (Investigations) | NA | NA | 14 (29)
Cytokine release syndrome (Immune system disorders) | NA | NA | 2
Dehydration (Metabolism and nutrition disorders) | NA | NA | 2 (4)
Depression (Psychiatric disorders) | NA | NA | 4 (5)
Diarrhea (Gastrointestinal disorders) | NA | NA | 15 (27)
Dizziness (Nervous system disorders) | NA | NA | 8 (11)
Dry Eye (Eye disorders) | NA | NA | 2
Dry Mouth (Gastrointestinal disorders) | NA | NA | 10 (10)
Dry skin (Skin and subcutaneous tissue disorders) | NA | NA | 5 (5)
Dysgeusia (Nervous system disorders) | NA | NA | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 6 (6)
Fullmess of ears (Ear and labyrinth disorders) | NA | NA | 2 (2)
Ear pain (Ear and labyrinth disorders) | NA | NA | 2 (2)
Edema limbs (General disorders) | NA | NA | 4 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | NA | NA | 2 (2)
TSH increased (Endocrine disorders) | NA | NA | 6 (8)
Elevated Free T4 (Endocrine disorders) | NA | NA | 3 (5)
Decreased TSH (Endocrine disorders) | NA | NA | 2 (2)
Low T4 (Endocrine disorders) | NA | NA | 3 (3)
Facial muscle weakness (Nervous system disorders) | NA | NA | 2 (2)
Fatigue (General disorders) | NA | NA | 25 (43)
Fever (General disorders) | NA | NA | 10 (18)
Flu like symptoms (General disorders) | NA | NA | 5 (7)
Gait disturbance (General disorders) | NA | NA | 2
Gastritis (Gastrointestinal disorders) | NA | NA | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | NA | NA | 4 (4)
Loose stools (Gastrointestinal disorders) | NA | NA | 6 (7)
Hemoptysis (Cardiac disorders) | NA | NA | 2
Hematoma (Vascular disorders) | NA | NA | 2 (2)
Genrealized muscle weakmess (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (5)
Headache (Nervous system disorders) | NA | NA | 18 (25)
Hypercalcemia (Metabolism and nutrition disorders) | NA | NA | 7 (8)
Hyperglycemia (Metabolism and nutrition disorders) | NA | NA | 25 (67)
Hyperkalemia (Metabolism and nutrition disorders) | NA | NA | 4 (6)
Hypertension (Vascular disorders) | NA | NA | 10 (20)
Hyperthyrodism (Endocrine disorders) | NA | NA | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | NA | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | NA | NA | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | NA | NA | 6 (10)
Hypokalemia (Metabolism and nutrition disorders) | NA | NA | 4 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | NA | NA | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | NA | NA | 18 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | NA | NA | 4 (5)
Hypotension (Vascular disorders) | NA | NA | 2 (3)
Hypothyrodism (Endocrine disorders) | NA | NA | 12 (13)
Insomnia (Psychiatric disorders) | NA | NA | 7 (7)
INR Increased (Investigations) | NA | NA | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | NA | NA | 2 (2)
Localized Edema (General disorders) | NA | NA | 5 (5)
Lymphedema (Vascular disorders) | NA | NA | 10 (12)
Lymphocyte count decreased (Investigations) | NA | NA | 2 (5)
Malaise (General disorders) | NA | NA | 2 (2)
Mucositis (Oral) (Gastrointestinal disorders) | NA | NA | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | 8 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | NA | NA | 12 (13)
Nausea (Gastrointestinal disorders) | NA | NA | 17 (27)
Neck edema (General disorders) | NA | NA | 2 (2)
Neck pain (General disorders) | NA | NA | 2 (2)
Neutorphil count decreased (Investigations) | NA | NA | 2 (2)
Non-cardiac chest pain (Cardiac disorders) | NA | NA | 4 (6)
Pain (General disorders) | NA | NA | 16 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | NA | 8 (9)
Papulopustular rash (Infections and infestations) | NA | NA | 2 (4)
Paresthesia (Nervous system disorders) | NA | NA | 7 (8)
Peripheral motor neuropathy (Nervous system disorders) | NA | NA | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | NA | NA | 5 (7)
Platelet count decreased (Investigations) | NA | NA | 5 (5)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | NA | NA | 21 (29)
Rash acneiform (Skin and subcutaneous tissue disorders) | NA | NA | 4 (5)
Rash maculo-papular (General disorders) | NA | NA | 19 (32)
Sinusitis (Infections and infestations) | NA | NA | 5 (5)
Vitiligo (Skin and subcutaneous tissue disorders) | NA | NA | 3 (4)
Sking Hypopigmentation (Skin and subcutaneous tissue disorders) | NA | NA | 5 (7)
Skin Infection (Infections and infestations) | NA | NA | 8 (17)
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | 6 (6)
Syncope (Nervous system disorders) | NA | NA | 2 (2)
Thromboembolic event (Vascular disorders) | NA | NA | 2 (2)
Tinnitus (Ear and labyrinth disorders) | NA | NA | 2 (2)
Toothache (Gastrointestinal disorders) | NA | NA | 2 (2)
Urinary Tract infection (Renal and urinary disorders) | NA | NA | 3 (3)
Vertigo (Ear and labyrinth disorders) | NA | NA | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2 (2)
Vomiting (Gastrointestinal disorders) | NA | NA | 10 (14)
Weight Loss (Investigations) | NA | NA | 4 (6)
White blood cell decreased (Blood and lymphatic system disorders) | NA | NA | 7 (18)
Wound complication (Injury, poisoning and procedural complications) | NA | NA | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | NA | NA | 2 (2)
Troponin I increased (Cardiac disorders) | NA | NA | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (2)
Sinus congestion (Congenital, familial and genetic disorders) | NA | NA | 4 (6)
Weakness to left eyelid (Eye disorders) | NA | NA | 2
Pain (bil eye lieds) (Eye disorders) | NA | NA | 2
Lower lid redness (Eye disorders) | NA | NA | 2
Photosensitivity (Eye disorders) | NA | NA | 2
Fecal incontinence (Gastrointestinal disorders) | NA | NA | 2
Fracture (Injury, poisoning and procedural complications) | NA | NA | 2
Gum infection (Gastrointestinal disorders) | NA | NA | 2
Hearing impaired (Ear and labyrinth disorders) | NA | NA | 2
Hemorrhoids (Gastrointestinal disorders) | NA | NA | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2
Ear infection (Infections and infestations) | NA | NA | 2
COVID-19 (Infections and infestations) | NA | NA | 3 (3)
Joint rang of motion decreased (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (4)
Lipase increased (Investigations) | NA | NA | 2
Lung Infections (Infections and infestations) | NA | NA | 2
Memory impairment (Nervous system disorders) | NA | NA | 2
Muscle weakness (left-sided) (Musculoskeletal and connective tissue disorders) | NA | NA | 2
Muscle weakness (lower limb) (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (2)
Muscle weakness-trunk (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (2)
Plantar fascitis (left foot) (Musculoskeletal and connective tissue disorders) | NA | NA | 2 (2)
Myocarditis (Cardiac disorders) | NA | NA | 2
Neurlgia (Nervous system disorders) | NA | NA | 2
Loose stools (Gastrointestinal disorders) | NA | NA | 6 (6)
Oral pain (Gastrointestinal disorders) | NA | NA | 2
Palpations (Cardiac disorders) | NA | NA | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2
Rectal hemorrhage (Renal and urinary disorders) | NA | NA | 2
Renal hemorrhage (Renal and urinary disorders) | NA | NA | 2
Sinus Bradycardia (Cardiac disorders) | NA | NA | 2
Sinus Tachycardia (Cardiac disorders) | NA | NA | 2
Soft tissue infection (Infections and infestations) | NA | NA | 2
Stomach pain (Gastrointestinal disorders) | NA | NA | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | NA | NA | 2
Tremor (Nervous system disorders) | NA | NA | 2
Upper respiratory infection (Infections and infestations) | NA | NA | 2
Uringary tract pain (Renal and urinary disorders) | NA | NA | 2
Weight gain (Investigations) | NA | NA | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | NA | NA | 2
Loose stools (Gastrointestinal disorders) | NA | NA | 7
Amnesia (Psychiatric disorders) | NA | NA | 2 (2)
Mood swings (Skin and subcutaneous tissue disorders) | NA | NA | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | NA | NA | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT02519322/Prot_SAP_000.pdf